CLINICAL TRIAL: NCT06965270
Title: Woman Mental Health and Addictions on Pregnancy
Acronym: WOMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Plan Nacional sobre Drogas (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015I073
Record Dates: First submitted 2025-03-20; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy; Mental Disorder; Substance Abuse
Keywords: Mental Health; Substance abuse; smoking; Dual disorders; Pregnancy
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders; Psychological Well-Being; Smoking | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment as usual (Active Comparator): Patients in this arm received the usual treatment provided by the health system
  Interventions: Behavioral: Treatment as usual
- Telematic intervention (Experimental): Patients in this arm received an App/internet-based psychotherapeutic intervention.
  Interventions: Behavioral: Internet/App intervention
- Standardized clinical intervention (Experimental): Patients in this arm received a standardized telephonic psychotherapeutic intervention.
  Interventions: Behavioral: Standardized clinical intervention

INTERVENTIONS:
Behavioral: Standardized clinical intervention — This manualized intervention consists of 8 sessions of evidence-based treatments for substance abuse and mental health problems.
  Session 1: Introduction, Psychoeducation, Assessment and Safety: Introduces what the patient's clinical assessment suggests about strengths and needs.
  Session 2: Relaxation, Mindfulness and cognitive distortions in CBT. Session 3: Getting started in Cognitive Restructuring (CR): thought challenge and action plan.
  Session 4: Craving management practice: includes challenging and replacing thoughts that lead to drug and alcohol use.
  Session 5: CR practice exercises and motivation: introduction to risk behaviors and triggers for drug and alcohol use. Relapse prevention.
  Session 6: Assertiveness and refusal techniques. Session 7: Problem solving, practice and reinforcement: CR skills, relaxation and relapse prevention applied in current circumstances.
  Session 8: Care plan and end of program.
  Arms: Standardized clinical intervention
Behavioral: Internet/App intervention — Using an already developed Internet/App platform (MeMind), patients will have access to the same therapeutic components as in the standardized intervention arm, arranged in sessions by modules.
  Components will be released weekly and reminded via push notifications. Patients will also receive two counseling calls at weeks 1 and 8 to help with technical issues and review problems with the program modules.
  Arms: Telematic intervention
Behavioral: Treatment as usual — Patient will recieve the usual intervention provided by the Health system
  Arms: Treatment as usual

SUMMARY:
The study intend to achieve the following objectives

Objective 1: Develop a collaborative infrastructure among different hospital services to support research that improves the accessibility, quality, and outcomes of integrated mental health services for pregnant women for tobacco, benzodiazepine, and other substance use and/or mental health problems.

Objective 2: To evaluate the effect and test the application of computer/smart phone based tools that can assist in the goal of achieving broader effect, improved accessibility and outcomes of substance abuse/mental health services in at-risk populations.

Objective 3: Conduct research on mental health services that: (a) emphasize rapid screening and referral; (b) test the feasibility, acceptability, and effectiveness of two different comprehensive behavioral treatment approaches (standardized clinical intervention and smart phone/computer-based intervention) for pregnant women with tobacco, benzodiazepine, and other substance use problems and mental health disorders; and (c) measure and decrease the obstetric, pediatric, and mental health consequences of these problems on the mother and child.

To achieve these objectives, investigators propose a system of evaluation and recruitment of patients in five Gynecology Departments that annually attend 3700 deliveries. A telematic intervention system based on a platform that we have used for other studies (Memind) and finally a randomized blinded clinical trial of 3 branches with 100 patients per branch (usual treatment, telematic intervention and standardized clinical intervention).

ELIGIBILITY:
Inclusion criteria:

1. Two or more positive responses to the AC-OK-Mental Health (AC-OK MH)subscale AND
2. One or more positive responses to the AC-OK-Substance Abuse (AC-OK SA) subscale and/or reported smoking more than once a month AND
3. No use of specialized services, defined as not having an appointment in the following month and have not seen a clinician in the past three months and
4. if the Paykel Suicide Scale was administered, they answered NO to questions 4 and 5.

Exclusion criteria:

1. Had received a diagnosis of psychotic or bipolar-related disorders or
2. Lacked capacity to consent, as determined by not being able to answer questions of the study purpose or process.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2014 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Depression symptoms | 12 months after enrollment
  Changes in the following scale were measured at 2,4,8,and 12 months:
  - Patient Health Questionnaire (PHQ-9) which addresses the nine DSM-IV diagnostic criteria for major depressive disorder. The range of scores goes from 0 to 27 points depending on the severity
Anxiety symptoms | 12 months after enrollment
  Changes in the following scale were measured at 2,4,8,and 12 months:
  - General Anxiety Disorder 7-item screener (GAD-7) for anxiety . The range of scores goes from 0 to 21 points depending on the severity
Post-Traumatic Stress Disorder symptoms | 12 months after enrollment
  Changes in the following scale were measured at 2,4,8,and 12 months:
  - Post-Traumatic Stress Disorder Checklist (PCL-5), a self-report measure for the 17 DSM-IV symptoms of PTSD. Scores above 33 are considered at risk.
Alcohol Use Disorders | 12 months after enrollment
  Changes in the following scale were measured at 2,4,8,and 12 months:
  Alcohol Use Disorders Identification Test (AUDIT), a screener developed by the World Health Organization (WHO). Patients with scores greater than or equal to 3 are considered at risk.
Drug Abuse Disorders | 12 months after enrollment
  Changes in the following scale were measured at 2,4,8,and 12 months:
  Drug Abuse Screening Test (DAST), a brief self-report instrument designed for drug abuse and dependence disorders detection. Patients with scores greater than or equal to 3 are considered at risk.
Smoking Dependence | 12 months after enrollment
  Changes in the following scale were measured at 2,4,8,and 12 months:
  Fagerström Test for Nicotine Dependence: A six item instrument that evaluates the amount of cigarette consumption, compulsion to smoke, and smoking dependence. The range of scores goes from 0 to 10 points depending on the dependence degree.
Substance use intensity | 12 months after enrollment
  At 2,4,8,and 12 months, women were asked about the number of days in the last month they used the following substances: alcohol, opioids, barbiturates, benzodiazepines, cocaine, amphetamines, cannabis, hallucinogens and inhalants

SECONDARY OUTCOMES:
Obstetric outcomes (Gestational week at birth) | 12 months after enrollment
  After birth, we measured the gestational week at the time of birth (number of weeks)
Obstetric outcomes (route of delivery) | 12 months after enrollment
  After birth, we evaluated the route of delivery (euthocic vaginal or instrumental delivery or cesarean section) and the reason for the indication of cesarean section.
Obstetric outcomes (puerperal complications ) | 12 months after enrollment
  After birth, we evaluated the presence of puerperal complications (Yes/no)
Child Perinatal outcomes (Fetal birth weight) | 12 months after enrollment
  After birth, we measured fetal birth weight (gr)
Child Perinatal outcomes (Apgar score) | 12 months after enrollment
  After birth, we measured Apgar score, assessed at one and five minutes.
Child Perinatal outcomes (Arterial pH) | 12 months after enrollment
  After birth, we measured Arterial pH
Child Perinatal outcomes (resuscitation) | 12 months after enrollment
  After birth, we measured the Need (Yes/no) and type of resuscitation (0-V)

IPD SHARING:
Plan to Share IPD: Yes